CLINICAL TRIAL: NCT05257694
Title: A Deep Learning Model Based on Contrast-enhanced Ultrasound to Aid Clinical Decisions and Predict Biological Biomarker and Prognosis of Hepatocellular Carcinoma
Brief Title: Clinical Decision Biological Biomarker and Prognosis Prediction of Hepatocellular Carcinoma by Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ping Liang (Other)
Responsible Party: Sponsor-Investigator, Ping Liang, Chief of department of interventional ultrasound, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2022-002
Record Dates: First submitted 2022-02-13; First posted 2022-02-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma; Contrast-enhanced Ultrasound; Prognosis; Surgery; Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — hepatectomy
Procedure: Ablation (Microwave ablation or Radiofrequency ablation) — image-guided ablation

SUMMARY:
Developing a deep learning model based on contrast-enhanced ultrasound (CEUS) to predict the prognosis of hepatocellular carcinoma (HCC) and aid choose operation decisions

DETAILED DESCRIPTION:
Collecting CEUS and clinical data of HCC from different institutions retrospectively.

Developing a deep learning model based on CEUS to predict the prognosis of HCC. Developing a deep learning model based on CEUS to choose a better operation (ablation or surgery) of HCC patients.

Then, validating the deep learning model in the prospective data.

ELIGIBILITY:
Inclusion Criteria:

* patients with HCC (Ia, Ib, IIa stage) China liver cancer staging who underwent resection or ablation
* without macro-vascular invasion
* Child-Pugh A/B grade
* HCC is proved by pathological examination or two enhanced imaging
* CEUS (Sonovue or Sonozoid) images are performed two weeks before the operation
* Invasive biomarker or prognosis of HCC available
* CEUS images are included in at least three stages (Arterial phase, Portal phase, and Late phase)

Exclusion Criteria:

* postop follow-up loss or expired less than 3 months
* patients with co-malignancy
* poor images quality for analyzing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HCC corresponding to Ia, Ib, IIa stage (China liver cancer staging) who undergo resection or ablation.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Immediately after the surgery or ablation
  Recurrence-free survival is defined as the time elapsed between a predefined point in time (the date of diagnosis, randomization or the intervention) and any recurrence (local, regional, or distant) or death due to any cause (death is an event).

SECONDARY OUTCOMES:
Recurrence | Immediately after the surgery or ablation
  Recurrence included local tumor progression, regional recurrence, or distant recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China